CLINICAL TRIAL: NCT02201550
Title: Regulation of Immune Cells in Obese Patients With Type 2 Diabetes Mellitus Treated With Liraglutide (Victoza)
Brief Title: Study of Immune Cells in Obese Patients With Type 2 Diabetes Mellitus Treated With Liraglutide
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Zealand Pharma (Industry)
Responsible Party: Principal Investigator, Carsten Dirksen, MD, PhD, Hvidovre University Hospital
Other Study IDs: H-2-2012-148-KLB
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liraglutide: Patients with type 2 diabetes undertaking treatment with liraglutide

SUMMARY:
The purpose of this study is to determine the effect of exogenous glucagon-like peptide-1 on the immune system i.e on the regulation of immune cells important in diseases such as obesity and diabetes.

The hypotheses are:

* Glucagon-like peptide-1 has an immunological effect observed by studying immune cells in the blood
* Treatment with glucagon-like peptide-1 increases the number of immune cells in the blood
* Treatment with glucagon-like peptide-1 leads to a more anti-inflammatory cytokine profile in the blood

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* BMI > 27 kg/m2
* Planed start of treatment with liraglutide
* Age > 18 years

Exclusion Criteria:

* Infection or active inflammatory disorder
* Immunomodulating treatment (i.e nonsteroidal antiinflammatory drugs, glucocorticoids)
* Smoking
* Alcohol consumption > 14 beverages/week
* Former bariatric surgery

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes undertaking treatment with liraglutide
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in number of specific immune cells in blood detected by flow cytometry | Before and 12 weeks after initiation of liraglutide treatment

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Dirksen, MD, PhD, Principal Investigator — Hvidovre University Hospital; Sten Madsbad, MD, DMSc, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark